CLINICAL TRIAL: NCT06272682
Title: Systemic Versus Local Corticosteroids in the Treatment of Carpal Tunnel Syndrome. Prospective Randomised Controlled Non-inferiority Study.
Brief Title: Corticosteroids in Carpal Tunnel Syndrome. Prospective Randomised Controlled Non-inferiority Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Jorge Guillermo Boretto, Principal Investigator, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6669
Record Dates: First submitted 2024-02-05; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: clinical trial; corticosteroid infiltration; carpal tunnel syndrome; betamethasone
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, controlled, non-inferiority analytical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Branch A: Local corticosteroid infiltration under ultrasound (Experimental): One dose. 1 ml Betamethasone acetate 6mg/2ml + Betamethasone disodium phosphate 6mg/2ml
  Interventions: Procedure: Local bethametasone injection
- Branch B: treated with intramuscular corticosteroid injection (Experimental): One dose. 2 ml Betamethasone acetate 6mg/2ml + Betamethasone disodium phosphate 6m/2ml.
  Interventions: Procedure: Systemic bethametasone injection

INTERVENTIONS:
Procedure: Systemic bethametasone injection — betamethasone intramuscular injection in the treatment of carpal tunnel syndrome
  Arms: Branch B: treated with intramuscular corticosteroid injection
Procedure: Local bethametasone injection — Local betamethasone injection under ultrasound in the carpal tunnel, in the treatment of carpal tunnel syndrome
  Arms: Branch A: Local corticosteroid infiltration under ultrasound

SUMMARY:
The goal of this prospective, randomised, controlled, non-inferiority analytical study is to compare the Boston score in patients treated with systemic (intramuscular) versus local infiltration corticosteroids in mild and moderate carpal tunnel syndrome in patients over 18 years of age with mild or moderate carpal tunnel syndrome.

The main questions it aims to answer are:

* What is the effectiveness of intramuscular injection of corticosteroids compared to local infiltration in the treatment of mild/moderate carpal tunnel syndrome?
* What are the adverse effects and application site pain associated with each route of administration?

Patients who meet the inclusion criteria will be asked to participate in the study and sign an informed consent form.

The Redcap randomizer will be used to assign the patient to one of the branches.

Researchers will compare

* Branch A: patients treated with local corticosteroid infiltration in carpal tunnel under ultrasound
* Branch B: patients treated with intramuscular corticosteroid injection.

Researchers will:

* Compare Boston Carpal Tunnel Questionnaire score at 1.5 months, 3 months, 6 months and 12 months post-procedure.
* Describe adverse reactions associated with the route of administration.
* Compare the pain at the site of application associated with the route of administration.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common peripheral compressive neuropathy of the upper limb, consisting of involvement of the median nerve at the level of the carpal tunnel. It has a prevalence of 7% to 16% in the United Kingdom adult population, while in the United States between 400/500 thousand patients are treated surgically, with an annual economic cost exceeding $2 billion.

A variety of treatments are available according to the stage of the pathology, including splinting, kinesic therapy, ultrasound, non-steroidal anti-inflammatory drugs, systemic or local corticosteroids , as well as surgical treatment in patients who do not respond to previous options.

Corticosteroid infiltration is one of the most widely used methods for the treatment of idiopathic carpal tunnel syndrome (ICTS) in mild and moderate stages, and short-term symptomatic improvement is reported in the literature, although the optimal dose and drug used for the same is varied in the various published studies, and is still a matter of debate in the literature. Betamethasone has greater anti-inflammatory power and a longer duration of action at the same equivalent dose than other corticosteroids used in the treatment of CTS (prednisolone, methylprednisolone, triamcinolone, cortisone).

In addition, ultrasound-guided local infiltration helps prevent iatrogenic injury compared to anatomical repair-guided infiltration. Studies show improvement in scores assessing symptomatology, although there is no strength in determining improvement in functional and electromyographic assessment. The rate of adverse reactions with this technique is low, reported to be <0.1% for major complications, and 2% for minor complications.

The effectiveness of local and systemic corticosteroids has been demonstrated, but whether there is any difference in clinical improvement in patients between one route of administration versus the other remains a question mark.

Rationale for the study In the institution, both intramuscular and ultrasound-guided administration of systemic corticosteroids are part of standard practice, with systemic administration indicated in the trauma department and ultrasound-guided administration in the rheumatology department. Although, given that these are standard practices, retrospective evaluation of the cases could answer the objective of this study, in the review of the cases the investigators found an imbalance in the type of CTS in the cohorts treated in each department. This is mainly due to the fact that in the orthopaedics service most patients consult for CTS and in the rheumatology service, due to the speciality itself, there is a large proportion of patients with secondary CTS (rheumatoid arthritis, juvenile arthritis, gout, etc.). Because of this, and to avoid patient selection bias, the aim of this study was to compare the efficacy of systemic (intramuscular) corticosteroid treatment with local infiltration in ICTS.

The same efficacy of systemic administration (intramuscular) as local administration (via ultrasound-guided infiltration in the carpal tunnel) should reduce the cost of treatment and the complications associated with local injection. In addition, it would allow effective treatment in centres where there are no specialists trained in the ultrasound-guided infiltration technique, allowing greater generalization of the treatment.

The investigator's hypothesis is that intramuscular corticosteroid infiltration (systemic effect) offers the same results in terms of symptom improvement as locally applied corticosteroids under ultrasound.

The primary objective is to compare the Boston score in patients treated with systemic (intramuscular) versus local infiltration corticosteroids in mild and moderate ICTS at 1.5 months, 3 months, 6 months and 12 months post-procedure.

The exploratory objectives are to describe adverse reactions associated with the route of administration and to compare the pain at the site of application associated with both methods, in relation to the technique used, measured with the Visual Analogue Pain Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Clinical diagnosis of mild/moderate idiopathic Carpal Tunnel Syndrome (paresthesias in the territory of the median nerve: in fingers 1, 2, 3 and radial border of 4 of the hand, nocturnal hand pain, and Positive Tinel's test, or Positive Phalen's test, or Positive Durkan's test)
* Diagnosis by electromyography and sensory and motor conduction velocity of mild/moderate involvement
* Patients who have agreed to participate in the study and signed the informed consent form.

Exclusion Criteria:

* Cervical radiculopathy, polyneuropathy, brachial plexus pathologies, thoracic operculum syndrome
* Systemic diseases causing secondary Carpal Tunnel Syndrome (rheumatoid arthritis, diabetes with polyneuropathy, hypothyroidism with low adherence to treatment, chronic renal disease)
* Chronic corticosteroid therapy or regular use of non-steroidal anti-inflammatory drugs
* Severe carpal tunnel syndrome: signs of thenar atrophy, daytime pain, sensory deficit in median nerve territory (two-point discrimination test >10mm)
* Previous history of wrist or distal radius fracture
* Corticosteroid allergies
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-08-11 (Estimated); Study Completion 2025-10-11 (Estimated)

PRIMARY OUTCOMES:
Compare the Boston Carpal Tunnel Syndrome Questionnaire | 12 months
  Compare the Boston Carpal Tunnel Syndrome Questionnaire in patients treated with systemic (intramuscular) versus local infiltration corticosteroids
  Two scales:
  * Symptom severity scale (11 questions): sum of the score of each question divided by the number of questions, with the lower limit and lower severity1 , and the upper limit and higher severity 5
  * Functional status scale (8 questions): sum of the score of each question divided by the number of questions, with the lower limit and lower severity 1, and the upper limit and higher severity 5.

SECONDARY OUTCOMES:
Adverse reactions | 12 months
  To describe adverse reactions associated with the route of administration.
Pain at the site of application | 12 months
  To compare the pain at the site of application associated with both methods, in relation to the technique used
  Visual analogue scale for pain: subjective pain scale, from 0 as the lower limit to 10 as the upper limit, where 0 is "no pain" and 10 is "the worst possible pain".

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No
study that tries not to reveal the identity of the participants